CLINICAL TRIAL: NCT02322632
Title: An Open-label, Balanced, Randomized, Two-treatment, Two-sequence, Two-period, Single-dose, Crossover Oral Bioequivalence Study of Paricalcitol Capsules 4 mcg of Dr. Reddy's Laboratories Limited and Zemplar Capsules, 4 mcg of Abbott Laboratories, USA in Healthy, Adult, Human Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Paricalcitol Capsules, 4 mcg Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 280-01
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paricalcitol Capsules, 4 mcg (Experimental): Paricalcitol Capsules, 4 mcg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Paricalcitol Capsules, 4 mcg
- Zemplar Capsules, 4 mcg (Experimental): Zemplar Capsules, 4 mcg of Abott Laboratories USA
  Interventions: Drug: Paricalcitol Capsules, 4 mcg

INTERVENTIONS:
Drug: Paricalcitol Capsules, 4 mcg — Paricalcitol Capsules, 4 mcg of Dr. Reddy's Laboratories Limited
  Other Names: Zemplar

SUMMARY:
An open-label, balanced, randomized, two-treatment, two-sequence, two-period, single-dose, crossover oral bioequivalence study in healthy subjects under fasting conditions.

DETAILED DESCRIPTION:
An open-label, balanced, randomized, two-treatment, two-sequence, two-period, single-dose, crossover oral bioequivalence study of Paricalcitol Capsules 4 mcg of Dr. Reddy's Laboratories Limited and Zemplar® Capsules 4 mcg of Abbott Laboratories, USA in healthy, adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, human volunteers between 18 and 55 years of age (both inclusive) living in and around Ahmedabad city of western part of India.
* Having a Body Mass Index (BMI) between 18.5 and 24.9 (both inclusive), calculated as weight in kg/height in m2.
* Have no significant diseases or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12- lead ECG and X-ray chest (postero-anterior view) recordings.
* Volunteers who have normal calcium, phosphorous status and no hypertensive status in order to avoid effect on vitamin D concentration in blood.
* Able to comply with the study procedures, in the opinion of the Principal investigator.
* Able to give voluntary informed consent for participation in the trial.

In case of female subjects*:

* Surgically sterilized at least 6 months prior to study participation; Or
* If of child bearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study.
* Urine pregnancy test (for female subjects*) must be negative at the time of screening. *No female subjects were enrolled in the study.

Exclusion Criteria:

* Known hypersensitivity or idiosyncratic reaction to Paricalcitol or to any of its excipients or any drug or any substance.
* History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
* Ingestion or Use of any medication at any time in 14 days prior to dosing. In any such case subject selection will be at the discretion of the Principal Investigator.
* Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAID induced urticaria.
* Consumption of Grapefruits or its products within a period of 48 hours prior to check-in.
* A recent history of harmful use of alcohol(less than 2 years), i.e. alcohol consumption of more than 14 standard drinks per week for men and more than 7 standard drinks per week for women (A standard drink is defined as 360 ml of beer or 150 ml of wine or 45 ml of 40% distilled spirits, such as rum, whisky, brandy etc). " or consumption of alcohol or alcoholic products within 48 hous prior to check-in.
* Smokers, who smoke 10 or more than 10 cigarettes / day or inability to abstain from smoking during the study.
* The presence of clinically significant abnormal laboratory values during screening.
* Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.
* History or presence of psychiatric disorders.
* A history of difficulty with donating blood.
* Donation of blood (1 unit or 350 mL) or receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication. Elimination half-life of the study drug should be taken into consideration for inclusion of the subject in the study. Note: In case the blood loss is ≤ 200 mL, subject may be enrolled 60 days after blood donation or last sample of the previous study.
* A positive hepatitis screen including hepatitis B surface antigen and anti- HCV antibodies.
* A positive test result for anti-HIV antibody.
* An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the study drug and throughout the subjects' participation in the study. In any such case subject selection will be at the discretion of the Principal Investigator. Nursing mothers (females)*. *No female subjects were enrolled in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Area under curve | 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36.0, 48.0 and 60.0 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Pankaj Kumar Jha, MD, Principal Investigator — Lambda Therapeutic Research Limited
Locations (1):
- Lambda Therapeutic Research Ltd, Ahmedabad, Gujarat, India